CLINICAL TRIAL: NCT05230160
Title: Can Intermittent Fasting Induce Weight Loss and Improve Gut Health as Compared to Standard Medical Care in Patients With Obesity/High BMI and Crohn's Disease.
Acronym: CD-Fast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Maitreyi Raman, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB21-1539
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The IF group will fast for 16 consecutive hours on 6 days per week with an 8-hour eating window (e.g., eat from 10 a.m. to 6 p.m.). The IF group will consume their habitual diet in terms of food choices and energy intake, but only during the 8-hour and full-day non-fasting periods. An RD will meet virtually with participants in the IF group at baseline to teach them the fasting protocol and how to manage energy intake and hunger, as well as to reinforce the requirement to not change habitual dietary practices. The research coordinator will call patients every two weeks to assess for changes in medications, compliance with the fasting protocol, and symptoms (assessed monthly) using the modified HBI.
  Interventions: Other: Intermittent Fasting
- Standard Medical Care Group (No Intervention): The control group will continue with their habitual dietary pattern. The research coordinator will call patients at baseline and every two weeks to assess for changes in medications and symptoms (assessed monthly) using the modified HBI.

INTERVENTIONS:
Other: Intermittent Fasting — Intermittent Fasting (IF) is a dietary intervention that involves periodic intervals of no or very limited energy intake. Fasting and feeding intervals vary and the practice of IF commonly consists of either a daily fast for 16 hours, a 24-hour fast on alternate days, or a fast two days per week on non-consecutive days.
  For the study, the IF group will be asked to fast for 16 consecutive hours, 6 days per week. This means they will have an 8-hour eating window (e.g., eat from 10 a.m. to 6 p.m.) each day. They will be asked to eat the same types of food and the same amounts as usual, but only during the 8-hour eating window.
  Arms: Intervention Group

SUMMARY:
Diet is a determinant of gut microbial diversity and composition and is recognized as a potential environmental trigger for IBD; for example, high-fat diets are associated with increased risk of CD in pre-clinical models, with effects mediated through dysbiosis and altered gut permeability.

Diet is also a potential non-pharmacological therapy for weight loss and for reducing the occurrence of disease flares and the reliance on dose escalation of biologic agents. Indeed, there is accumulating evidence for the role of diet in the treatment of CD, and diet-induced improvement of microbial dysbiosis is associated with induction of remission in pediatric patients with active CD.

Intermittent Fasting (IF) is a dietary intervention that involves periodic intervals of no or very limited energy intake. We want to determine the efficacy and feasibility of a 12-week IF(Intermittent Fasting) intervention to induce weight loss (by 1 BMI unit reduction), decrease biomarker inflammation and increase microbial functional diversity compared to standard medical management (SM) in a pilot study of individuals with overweight or obesity and CD in clinical remission with elevated biomarkers of inflammation, indicated by fecal calprotectin (FCP) > 250 µg/g or C-reactive protein (CRP) > 5 mg/L).

DETAILED DESCRIPTION:
Objectives: To determine if a 12-week IF intervention compared to SM:

1. Induces weight loss of at least 1 BMI unit.
2. Reduces intestinal and systemic inflammation.
3. Alters gut microbial community structure (beta-diversity) from baseline.
4. Alters the adipokines and myokines leptin, adiponectin, IL-6, or irisin.
5. Alters zonulin and serum levels of gastrointestinal hormones ghrehlin, glucagon-like peptide 1 (GLP-1), and glucagon-like peptide 2 (GLP-2).
6. Alters body composition and whether changes in body composition have an effect on biomarkers of inflammation.
7. Is a feasible and sustainable intervention for patients with CD.

Hypotheses: We hypothesize that, compared to SM, IF will:

1. Induce at least a 1-unit decrease in BMI over the course of the intervention.
2. Improve inflammatory markers of CD, demonstrated by a decrease in FCP by ≥ 50%, normalization of FCP to ≤ 100 µg/g, or a decrease in CRP to ≤ 5 mg/L.
3. Alter gut microbial community structure (beta-diversity ) and lead to enrichment of bacterial species typically depleted in CD, such as Faecalibacterium prausnitzii and Roseburia hominus with concomitant decreases in Escherichia coli and overall Proteobacteria phylum abundance.
4. Alter adipokines and myokines (leptin, adiponectin, IL-6, and irisin), zonulin and serum levels of gastrointestinal hormones (ghrehlin, GLP-1, and GLP-2).
5. Alter body composition by decreasing VAT.
6. Be a feasible and sustainable treatment option for patients with CD

Methods

Study Design:

The study is a 12-week pilot randomized controlled trial (RCT). Eligible participants (N=42) will be randomized 1:1 to either the IF or the SM control group. Patients from the University of Calgary IBD clinic will be enrolled in the RCT.

Screening:

The study RD will assess participants for malnutrition using the abridged patient-generated subjective global assessment (PG-SGA), a validated tool to determine malnutrition status in patients with chronic disease. The Nine Item Avoidant/Restrictive Food Intake Disorder screen33 will be completed to rule out avoidant and restrictive food behaviours that may increase the malnutrition risk of an IF intervention.

Inclusion criteria:

1) ≥ 18 to ≤ 75 years of age; 2) ileocolonic or colonic CD in clinical remission diagnosed through conventional definitions with a Harvey Bradshaw Index (HBI) < 5 within 3 months of recruitment; 3) presence of inflammation using an FCP ≥ 250 µg/g or a CRP ≥ 5 mg/L; 4) stable dosing of biologic agents and/or immunomodulators and/or oral or rectal 5-ASA, and no changes to medical management (including corticosteroid exposure) for at least 3 months prior to recruitment; and 5) presence of overweight or obesity with BMI > 25 and a PG-SGA of class A.

Exclusion criteria:

1) upper gastrointestinal involvement CD, fistulizing disease; 2) documented strictures based on sonographic findings or colonoscopy within the last year; 3) > 1 small bowel resection; 4) colectomy; 5) presence of an ostomy; 6) antibiotic use in past 3-months; 7) pregnancy; and 8) corticosteroids in the last 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 to ≤ 75 years of age;
2. ileocolonic or colonic CD in clinical remission diagnosed through conventional definitions with a Harvey Bradshaw Index (HBI) < 5 within 3 months of recruitment;
3. presence of inflammation using an FCP ≥ 250 µg/g or a CRP ≥ 5 mg/L;
4. stable dosing of biologic agents and/or immunomodulators and/or oral or rectal 5-ASA, and no changes to medical management (including corticosteroid exposure) for at least 3 months prior to recruitment
5. presence of overweight or obesity with BMI > 25 and a PG-SGA of class A.

Exclusion Criteria:

1. upper gastrointestinal involvement CD, fistulizing disease;
2. documented strictures based on sonographic findings or colonoscopy within the last year;
3. > 1 small bowel resection;
4. colectomy;
5. presence of an ostomy;
6. antibiotic use in past 3-months;
7. pregnancy;
8. corticosteroids in the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
BMI-A decrease in BMI of at least 1 BMI unit over the course of the intervention: Change is being assessed | Baseline and Week 12
  A measure of body fat based on height and weight
Fecal Calprotectin: Change is being assessed | Baseline and Week 12
  FCP is a test used to detect inflammation in the colon and is associated with disease
C Reactive Protien: Change is being assessed | Baseline and Week 12
  A protein the liver produces in the presence of inflammatory disease

SECONDARY OUTCOMES:
24 hour ASA food recalls: Change is being assessed. | Baseline and week 12
  Assess diet quality
Serum and fecal metabolomics: Change is being assessed | Baseline and Week 12
  Metabolomics analysis provides a snapshot of an organism's current metabolite profile
Serum markers: Change is being assessed | Baseline and week 12
  Leptin, adiponectin, IL-6, irisin, zonulin, ghrehlin, GLP-1, and GLP-2
Body Composition: Change is being assessed | Baseline and week 12
  Lean muscle mass, total fat mass, subcutaneous fat mass, and visceral fat mass will be assessed using DEXA, a gold standard test to determine body composition, differentiate proportion of lean muscle compared to fat mass, and distinguish between subcutaneous and VAT
Fecal microbiome: Change is being assessed | Baseline and Week 12
  Determined using shotgun metagenomic sequencing (Illumina NovaSeq 6000 platform at the UoC Centre for Health Genomics and Informatics) to provide in-depth coverage of the microbial metagenome. Sequences will be analyzed for species level abundances, beta diversity metrics, and functional capacity based on gene content.

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Raman, MD, Principal Investigator — University of Calgary
Locations (1):
- TRW building, Foothills, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No There is no plan to make individual participant data available to other researchers outside of the study team.